CLINICAL TRIAL: NCT04944251
Title: Exercise in Persons With Multiple Sclerosis
Brief Title: Regular Exercise Improves Physical Capacity and Promotes Neurotrophins in Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Mehmet Acik, Principal Investigator,, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19-4T/43
Record Dates: First submitted 2021-05-20; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Multiple Sclerosis; Exercise Intervention; Neuro-Degenerative Disease
Keywords: multiple sclerosis; exercise; nerve growth factor; neurotrophin 3; cognition; quality of life
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity; Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Intervention Model Description: randomized prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- aerobic exercise group (Experimental): the patients in the aerobic group started to exercise at a heart rate corresponding to 60% of the maximal VO2, by adjusting the pedal resistance of the exercise bike, consistent with the Karvonen formula. This was followed by exercise cycling at a heart rate corresponding to 70% of maximal VO2 in the second month, and 80% of maximal VO2 in the third month, for 30 minutes, 3 days a week
  Interventions: Behavioral: Regular Exercise
- strength exercise group (Experimental): The patients included in the strength exercise group performed weight training exercises involving 10 large muscle groups (leg press, chest press, leg curl, lateral pull down, leg extension, dumbbell lateral raise, calf press, upright row, sit up, quadruped arm opposite leg raise), 3 days a week; including 1 set of 12-15 repetitions in the first month, 2 sets of 12-15 repetitions in the second month, and 3 sets of 12-15 repetitions in the third month (Figure 1). Participants' working weights were set as 60% of the maximum weight they could lift.
  Interventions: Behavioral: Regular Exercise
- control group (No Intervention): The patients who didn't want to exercise were included in the control group.

INTERVENTIONS:
Behavioral: Regular Exercise — the third month, for 30 minutes or 1 hour, 3 days a week
  Arms: aerobic exercise group; strength exercise group

SUMMARY:
ABSTRACT

Objective:

The investigators aimed to determine the effect of regular exercise on aerobic capacity, strength values, and plasma levels of nerve growth factor (NGF) and Neurotrophin-3 (NT-3) in patients with multiple sclerosis (MS), and investigate its effects on MS symptoms including cognitive impairment, fatigue, balance disorders and quality of life.

Methods:

Forty-three relapsing-remitting MS (RRMS) patients with an EDSS score of 4 or less participated in the study. Participants were divided into 3 groups as aerobic exercise, strength exercise and control groups. The patients in the exercise groups had exercise programs 3 days a week, for 3 months. Aerobic capacity (maximum VO2 value), strength measurements and balance tests were done, and NGF and NT-3 plasma levels were analyzed in all participants at the beginning and end of the study. MSQoL54 quality of life, fatigue impact scale (FIS), Pittsburgh Sleep Quality Index (PSQI) and BICAMS scale were applied to evaluate cognitive functions.

DETAILED DESCRIPTION:
INTRODUCTION Multiple sclerosis (MS) is a chronic inflammatory and neurodegenerative disorder characterized by inflammation, demyelination, axonal damage and gliosis, particularly affecting white matter, and also gray matter 1. It is the most common disorder of the central nervous system (CNS) that causes neurological disability in young adults. Various degrees of physical and cognitive impairments are seen starting in the early period, and particularly in the progressive course of the disease 2.

Physical inactivity may lead to progressive muscle atrophy in MS patients due to insufficient neural stimulation to the muscles 6. In MS patients, maximal oxygen consumption (VO2 max), which is a marker of cardiorespiratory fitness and functional performance, has been shown to decrease 7. All of these conditions may lead to worsening of MS symptoms and fatigue, which may result in a vicious cycle and cause reduced physical activity and an impairment in quality of life.

Exercise has numerous neurobiological effects, including anatomical and physiological changes in the brains of healthy and unhealthy individuals 8. Exercise provides comprehensive alterations in cerebrovascular structures such as blood flow, nutrient delivery, development of angiogenesis and regeneration of blood vessels 9. These alterations facilitate neurogenesis, increase synaptic plasticity, and ultimately may improve brain health and MS-related symptoms 9. Neurotrophins (NT) are growth factors that provide the survival and hypertrophy of neurons, as well as neurogenesis and synaptic plasticity 10. They are synthesized by a number of cell types including peripheral nervous system neurons, peripheral tissues, and particularly in the CNS 11,12. It is believed that exercise activates molecules and cellular cascades that support and maintain brain plasticity, facilitates neurogenesis, and thus may be effective in neurodegenerative processes and cognitive disorders 13.

In this study, the investigators aimed to investigate the effect of regular exercise on aerobic capacity and strength values, and to determine whether exercise contributes to the improvement of cognitive, balance, and sleep disorders and fatigue, and quality of life in MS patients. The investigators also investigated post-exercise changes in the plasma levels of neurotrophins, nerve growth factor (NGF) and neurotrophin-3 (NT-3), which are important biomarkers in neural regeneration and re-myelination.

MATERIAL AND METHODS Study design A total of 53 relapsing remitting form MS (RRMS) patients between the ages of 18-55 years, diagnosed with definite MS according to 2017 McDonald criteria, and followed up in Ege University MS and Demyelinating Diseases Unit, without an MS attack in the last 3 months, had an EDSS score ≤ 4 that did not change with symptomatic or immunomodulatory treatments within 6 months were included in this prospective randomized controlled study. The procedures and possible side effects (such as exercise-related injuries and having an MS attack) were explained in detail to each participant candidate, and the "Informed Consent Form" was signed by the volunteers. "Ege University Clinical Research Ethics Committee" approved the study protocol (date: Apr 03, 2019, decree no: 19-4T/43).

The patients who participated in the study and wished to be included in the exercise group were randomly allocated to the aerobic exercise and strength exercise groups. The patients who didn't want to exercise were included in the control group. Four patients in the aerobic group and 6 patients in the strength group could not complete the study due to reasons such as knee pain (1), not attending exercise sessions regularly (8), and not attending control measurements (1).

Exercise Procedures:

The patients in the exercise groups carried out tailor-made exercise programs, under the supervision of a faculty member of the Faculty of Sports Sciences. It was paid attention to keep the temperature of the exercise room at 20°C. The control patients did not participate in any exercise or physical activity program.

In the first month, the patients in the aerobic group started to exercise at a heart rate corresponding to 60% of the maximal VO2, by adjusting the pedal resistance of the exercise bike, consistent with the Karvonen formula. This was followed by exercise cycling at a heart rate corresponding to 70% of maximal VO2 in the second month, and 80% of maximal VO2 in the third month, for 30 minutes, 3 days a week (Figure 1) 14.

The patients included in the strength exercise group performed weight training exercises involving 10 large muscle groups (leg press, chest press, leg curl, lateral pull down, leg extension, dumbbell lateral raise, calf press, upright row, sit up, quadruped arm opposite leg raise), 3 days a week; including 1 set of 12-15 repetitions in the first month, 2 sets of 12-15 repetitions in the second month, and 3 sets of 12-15 repetitions in the third month. Participants' working weights were set as 60% of the maximum weight they could lift.

ELIGIBILITY:
Inclusion Criteria:

* A total of 53 relapsing remitting form MS (RRMS) patients between the ages of 18-55 years, diagnosed with definite MS according to 2017 McDonald criteria, and followed up in Ege University MS and Demyelinating Diseases Unit, without an MS attack in the last 3 months, had an EDSS score ≤ 4 that did not change with symptomatic or immunomodulatory treatments within 6 months were included in this prospective randomized controlled study.

Exclusion Criteria:

* Patients who did not meet the inclusion criteria were excluded from the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-19 (Actual)

PRIMARY OUTCOMES:
Aerobic capacity assessment after exercise intervention | Each participant's progress will be tested at the beginning and end of the 12-week training period.
  Measurement of Aerobic Capacity: Milliliters were used for the amount of oxygen used, kilograms were used for body weight, and minutes were used for time. the amount of oxygen consumed, weight and time will be combined to report aerobic capacity in ml/kg/min.
  The unit of aerobic capacity, ml/kg/min, refers to the amount of oxygen the body consumes per kilogram per minute. The indirect Astrand test bicycle test protocol with Lode Corival bicycle ergometer was applied to all patients. The pedal resistance applied in the test and the mean pulse rate were marked in the Astrand normogram, and the aerobic capacities of the patients were calculated. It was observed that aerobic capacity (ml/kg/min) increased in exercise groups after regular exercise.
Strength assessment after exercise intervention | Each participant's progress will be tested at the beginning and end of the 12-week training period.
  Strength Measurements: The kilogram-force (kg-f) is a non-standard Gravitational Metric unit of force. The kilogram-force is equal to the magnitude of the force exerted on one kilogram of mass in a 9.80665 m/s2 gravitational field. Kilogram was used for weight. The force is any influence that, when unopposed, will change the motion of an object. Weight and force will be combined to report strength in kg-f. Strength was examined with an isometric hand and backleg dynamometer in all patients. Strength was examined with an isometric hand and backleg dynamometer in all patients. Two measurements were made, at the beginning and at the end of the study. It was observed that strength values increased in exercise groups after regular exercise.
plasma neurotrophin values (pg/ml) | Each participant's progress will be tested at the beginning and end of the 12-week training period.
  Plasma NGF and NT-3 levels were measured with an ELISA kit. Plasma neurotrophin values increased in exercise groups.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet ACIK, Dr, Principal Investigator — Ege University; Seckin Senisik, Ass. Prof., Study Director — Ege University; Nur Yuceyar, Professor, Study Director — Ege University
Locations (1):
- Ege University, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
For the continuity of scientific research, my data can be used for other researches.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: anyone who wishes to access the data.

REFERENCES:
- [Background] Lassmann H. Pathogenic Mechanisms Associated With Different Clinical Courses of Multiple Sclerosis. Front Immunol. 2019 Jan 10;9:3116. doi: 10.3389/fimmu.2018.03116. eCollection 2018. PMID 30687321
- [Background] Oh J, Vidal-Jordana A, Montalban X. Multiple sclerosis: clinical aspects. Curr Opin Neurol. 2018 Dec;31(6):752-759. doi: 10.1097/WCO.0000000000000622. PMID 30300239
- [Background] Bamer AM, Johnson KL, Amtmann D, Kraft GH. Prevalence of sleep problems in individuals with multiple sclerosis. Mult Scler. 2008 Sep;14(8):1127-30. doi: 10.1177/1352458508092807. Epub 2008 Jul 16. PMID 18632776
- [Background] Mazumder R, Murchison C, Bourdette D, Cameron M. Falls in people with multiple sclerosis compared with falls in healthy controls. PLoS One. 2014 Sep 25;9(9):e107620. doi: 10.1371/journal.pone.0107620. eCollection 2014. PMID 25254633
- [Background] Benedict RH, Wahlig E, Bakshi R, Fishman I, Munschauer F, Zivadinov R, Weinstock-Guttman B. Predicting quality of life in multiple sclerosis: accounting for physical disability, fatigue, cognition, mood disorder, personality, and behavior change. J Neurol Sci. 2005 Apr 15;231(1-2):29-34. doi: 10.1016/j.jns.2004.12.009. Epub 2005 Jan 26. PMID 15792817
- [Background] Jorgensen M, Dalgas U, Wens I, Hvid LG. Muscle strength and power in persons with multiple sclerosis - A systematic review and meta-analysis. J Neurol Sci. 2017 May 15;376:225-241. doi: 10.1016/j.jns.2017.03.022. Epub 2017 Mar 18. PMID 28431618
- [Background] Phillips C, Baktir MA, Srivatsan M, Salehi A. Neuroprotective effects of physical activity on the brain: a closer look at trophic factor signaling. Front Cell Neurosci. 2014 Jun 20;8:170. doi: 10.3389/fncel.2014.00170. eCollection 2014. PMID 24999318
- [Background] Lange-Asschenfeldt C, Kojda G. Alzheimer's disease, cerebrovascular dysfunction and the benefits of exercise: from vessels to neurons. Exp Gerontol. 2008 Jun;43(6):499-504. doi: 10.1016/j.exger.2008.04.002. Epub 2008 Apr 6. PMID 18474414
- [Background] Vilar M, Mira H. Regulation of Neurogenesis by Neurotrophins during Adulthood: Expected and Unexpected Roles. Front Neurosci. 2016 Feb 9;10:26. doi: 10.3389/fnins.2016.00026. eCollection 2016. PMID 26903794
- [Background] Riley CP, Cope TC, Buck CR. CNS neurotrophins are biologically active and expressed by multiple cell types. J Mol Histol. 2004 Nov;35(8-9):771-83. doi: 10.1007/s10735-004-0778-9. PMID 15609090
- [Background] Yamamoto M, Sobue G, Yamamoto K, Terao S, Mitsuma T. Expression of mRNAs for neurotrophic factors (NGF, BDNF, NT-3, and GDNF) and their receptors (p75NGFR, trkA, trkB, and trkC) in the adult human peripheral nervous system and nonneural tissues. Neurochem Res. 1996 Aug;21(8):929-38. doi: 10.1007/BF02532343. PMID 8895847
- [Background] Cotman CW, Berchtold NC. Exercise: a behavioral intervention to enhance brain health and plasticity. Trends Neurosci. 2002 Jun;25(6):295-301. doi: 10.1016/s0166-2236(02)02143-4. PMID 12086747
- [Background] KARVONEN MJ, KENTALA E, MUSTALA O. The effects of training on heart rate; a longitudinal study. Ann Med Exp Biol Fenn. 1957;35(3):307-15. No abstract available. PMID 13470504
- [Result] Langeskov-Christensen M, Heine M, Kwakkel G, Dalgas U. Aerobic capacity in persons with multiple sclerosis: a systematic review and meta-analysis. Sports Med. 2015 Jun;45(6):905-23. doi: 10.1007/s40279-015-0307-x. PMID 25739555
- [Result] Langeskov-Christensen M, Langeskov-Christensen D, Overgaard K, Moller AB, Dalgas U. Validity and reliability of VO(2)-max measurements in persons with multiple sclerosis. J Neurol Sci. 2014 Jul 15;342(1-2):79-87. doi: 10.1016/j.jns.2014.04.028. Epub 2014 Apr 27. PMID 24825731
- [Result] ASTRAND PO, RYHMING I. A nomogram for calculation of aerobic capacity (physical fitness) from pulse rate during sub-maximal work. J Appl Physiol. 1954 Sep;7(2):218-21. doi: 10.1152/jappl.1954.7.2.218. No abstract available. PMID 13211501
- [Result] Lippi G, Mattiuzzi C, Sanchis-Gomar F. Updated overview on interplay between physical exercise, neurotrophins, and cognitive function in humans. J Sport Health Sci. 2020 Jan;9(1):74-81. doi: 10.1016/j.jshs.2019.07.012. Epub 2019 Sep 6. PMID 31921482
- [Result] Ernfors P, Lee KF, Kucera J, Jaenisch R. Lack of neurotrophin-3 leads to deficiencies in the peripheral nervous system and loss of limb proprioceptive afferents. Cell. 1994 May 20;77(4):503-12. doi: 10.1016/0092-8674(94)90213-5. PMID 7514502
- [Result] Dominguez-Sanchez MA, Bustos-Cruz RH, Velasco-Orjuela GP, Quintero AP, Tordecilla-Sanders A, Correa-Bautista JE, Triana-Reina HR, Garcia-Hermoso A, Gonzalez-Ruiz K, Pena-Guzman CA, Hernandez E, Pena-Ibagon JC, Tellez-T LA, Izquierdo M, Ramirez-Velez R. Acute Effects of High Intensity, Resistance, or Combined Protocol on the Increase of Level of Neurotrophic Factors in Physically Inactive Overweight Adults: The BrainFit Study. Front Physiol. 2018 Jun 27;9:741. doi: 10.3389/fphys.2018.00741. eCollection 2018. PMID 29997519
- [Result] Manni L, Rocco ML, Bianchi P, Soligo M, Guaragna M, Barbaro SP, Aloe L. Nerve growth factor: basic studies and possible therapeutic applications. Growth Factors. 2013 Aug;31(4):115-22. doi: 10.3109/08977194.2013.804073. Epub 2013 Jun 19. PMID 23777359
- [Result] Briken S, Gold SM, Patra S, Vettorazzi E, Harbs D, Tallner A, Ketels G, Schulz KH, Heesen C. Effects of exercise on fitness and cognition in progressive MS: a randomized, controlled pilot trial. Mult Scler. 2014 Mar;20(3):382-90. doi: 10.1177/1352458513507358. Epub 2013 Oct 24. PMID 24158978
- [Result] Zheng F, Zhou X, Moon C, Wang H. Regulation of brain-derived neurotrophic factor expression in neurons. Int J Physiol Pathophysiol Pharmacol. 2012;4(4):188-200. Epub 2012 Dec 26. PMID 23320132
- [Result] Leavitt VM, Cirnigliaro C, Cohen A, Farag A, Brooks M, Wecht JM, Wylie GR, Chiaravalloti ND, DeLuca J, Sumowski JF. Aerobic exercise increases hippocampal volume and improves memory in multiple sclerosis: preliminary findings. Neurocase. 2014;20(6):695-7. doi: 10.1080/13554794.2013.841951. Epub 2013 Oct 4. PMID 24090098
- [Result] Frielingsdorf H, Simpson DR, Thal LJ, Pizzo DP. Nerve growth factor promotes survival of new neurons in the adult hippocampus. Neurobiol Dis. 2007 Apr;26(1):47-55. doi: 10.1016/j.nbd.2006.11.015. Epub 2006 Dec 20. PMID 17270453
- [Result] Erickson KI, Kramer AF. Aerobic exercise effects on cognitive and neural plasticity in older adults. Br J Sports Med. 2009 Jan;43(1):22-4. doi: 10.1136/bjsm.2008.052498. Epub 2008 Oct 16. No abstract available. PMID 18927158
- [Result] Paltamaa J, Sjogren T, Peurala SH, Heinonen A. Effects of physiotherapy interventions on balance in multiple sclerosis: a systematic review and meta-analysis of randomized controlled trials. J Rehabil Med. 2012 Oct;44(10):811-23. doi: 10.2340/16501977-1047. PMID 22990349
- [Result] Cakt BD, Nacir B, Genc H, Saracoglu M, Karagoz A, Erdem HR, Ergun U. Cycling progressive resistance training for people with multiple sclerosis: a randomized controlled study. Am J Phys Med Rehabil. 2010 Jun;89(6):446-57. doi: 10.1097/PHM.0b013e3181d3e71f. PMID 20216060
- [Result] Sadeghi Bahmani D, Kesselring J, Papadimitriou M, Bansi J, Puhse U, Gerber M, Shaygannejad V, Holsboer-Trachsler E, Brand S. In Patients With Multiple Sclerosis, Both Objective and Subjective Sleep, Depression, Fatigue, and Paresthesia Improved After 3 Weeks of Regular Exercise. Front Psychiatry. 2019 May 3;10:265. doi: 10.3389/fpsyt.2019.00265. eCollection 2019. PMID 31130879
- [Result] Yang PY, Ho KH, Chen HC, Chien MY. Exercise training improves sleep quality in middle-aged and older adults with sleep problems: a systematic review. J Physiother. 2012;58(3):157-63. doi: 10.1016/S1836-9553(12)70106-6. PMID 22884182
- [Result] Santos RV, Tufik S, De Mello MT. Exercise, sleep and cytokines: is there a relation? Sleep Med Rev. 2007 Jun;11(3):231-9. doi: 10.1016/j.smrv.2007.03.003. PMID 17517356
- [Result] Melancon MO, Lorrain D, Dionne IJ. Exercise and sleep in aging: emphasis on serotonin. Pathol Biol (Paris). 2014 Oct;62(5):276-83. doi: 10.1016/j.patbio.2014.07.004. Epub 2014 Aug 4. PMID 25104243
- [Result] Rooney S, Wood L, Moffat F, Paul L. Is Fatigue Associated With Aerobic Capacity and Muscle Strength in People With Multiple Sclerosis: A Systematic Review and Meta-analysis. Arch Phys Med Rehabil. 2019 Nov;100(11):2193-2204. doi: 10.1016/j.apmr.2019.06.014. Epub 2019 Aug 6. PMID 31398354
- [Result] Dalgas U, Stenager E, Jakobsen J, Petersen T, Hansen HJ, Knudsen C, Overgaard K, Ingemann-Hansen T. Fatigue, mood and quality of life improve in MS patients after progressive resistance training. Mult Scler. 2010 Apr;16(4):480-90. doi: 10.1177/1352458509360040. Epub 2010 Mar 1. PMID 20194584
- [Result] Motl RW, Snook EM. Physical activity, self-efficacy, and quality of life in multiple sclerosis. Ann Behav Med. 2008 Feb;35(1):111-5. doi: 10.1007/s12160-007-9006-7. Epub 2008 Feb 12. PMID 18347911
- See also: Results Reference — https://www.minervamedica.it/en/journals/medicina-dello-sport/article.php?cod=R26Y2016N02A0228
- See also: Results Reference — http://www.ijaep.com/index.php/IJAE/article/view/228